CLINICAL TRIAL: NCT00080587
Title: Atherosclerosis in the Coronary and Carotid Arteries: Correlations Between Coronary IVUS, Carotid Ultrasound, and Carotid MRI
Brief Title: Atherosclerosis in the Coronary and Carotid Arteries
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040154; 04-H-0154
Record Dates: First submitted 2004-04-07; First posted 2004-04-07 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-01

CONDITIONS: Coronary Disease
Keywords: Intravascular Ultrasound; Magnetic Resonance Imaging; Hyperlipidemia; Cholesterol; Coronary Artery Disease
MeSH Terms: conditions — Coronary Disease; Hyperlipidemias; Coronary Artery Disease

SUMMARY:
This study will compare changes in atherosclerotic plaque in the coronary arteries (vessels on the surface of the heart that supply blood to the heart) with changes in the carotid arteries (vessels in the neck that supply blood to the brain) in patients enrolled in a Pfizer-sponsored treatment trial for coronary artery disease. Atherosclerosis is a buildup of fatty deposits (plaque) in arteries that can lead to blockage of the vessel, possibly resulting in heart attack or stroke. A major question in cardiovascular disease is how closely atherosclerotic changes in the coronary arteries correlate with changes in the carotid artery that occur with treatment. substudy of a Pfizer.

Patients enrolled in the Pfizer trial comparing the effectiveness of the drug atorvastatin with a combination of atorvastatin and CETP inhibitor (a drug to increase HDL cholesterol levels) may be eligible for this substudy.

Participants undergo magnetic resonance imaging (MRI) and ultrasound of the carotid arteries to measure the thickness of the vessels. The results are then compared with the coronary artery images obtained as part of the patient's evaluation for the Pfizer trial.

MRI

MRI scans use a powerful magnet with an advanced computer system and radio waves to produce accurate, detailed pictures of organs and tissues. During the scan the patient lies on a table in a narrow cylinder containing a magnetic field, wearing earplugs to muffle loud noises that occur with electrical switching of the magnetic fields. A medicine called gadolinium contrast may be injected into a vein during part of the scan to brighten the images. The scan takes about 30 to 90 minutes. An electrocardiogram (ECG) is done during the scan to monitor the heart's electrical activity. Patients who agree to undergo another MRI test are also imaged in a scanner that uses a stronger (3 Tesla) magnet.

Ultrasound

An echocardiogram (ultrasound of the heart) uses sound waves to image the carotid arteries. A gel is applied to the area of the neck to be imaged and a small handheld ultrasound probe is held against the neck to take the pictures.

Participants return after 2 years for a second set of tests.

DETAILED DESCRIPTION:
Under the general hypothesis that atherosclerosis is a systemic disease; the purpose of this protocol is to compare coronary artery atherosclerotic abnormalities with carotid artery abnormalities. This is an NHLBI sponsored sub study to the Pfizer sponsored trial comparing atorvastatin or the combination of atorvastatin/CETP inhibitor as treatments for patients with coronary heart disease. The primary study is a multicenter, randomized, double blind, active-controlled study which uses intracoronary ultrasound to measure coronary plaque volume during the course of treatment. The scientific value of the NHLBI sub study will be the comparison of atherosclerotic abnormalities in two different vascular beds, the coronary artery and the carotid arteries. This study will examine correlations between invasive coronary measurements by intravascular ultrasound (IVUS), with 2-dimensional measurements of wall thickness by carotid intimal medial wall thickness (IMT), and with 3-dimensional measurements of carotid wall volume by MRI and 3D ultrasound. Secondary analysis will probe whether carotid plaque characteristics can predict atheroma regression. Secondary analysis will also assess the ability of noninvasive carotid measures to predict the degree of coronary regression determined in the coronary arteries by IVUS. It is important to note that the NHLBI study design remains blinded to the treatment group a subject is enrolled in since the sample size for a single center study is too small to detect the conservatively estimated additional benefit of combination atorvastatin/CETP inhibitor treatment over the already effective atorvastatin alone. Thus, the NHLBI sub study is primarily a pathophysiological study correlating carotid and coronary atherosclerotic changes as well as a technological comparison of IVU, carotid IMT, and carotid vessel wall volume by MRI. If successful, this study could provide the framework for following treatment trials of this nature with noninvasive tools, either ultrasound or MRI, in place of the accurate but invasive IVUS.

ELIGIBILITY:
INCLUSION CRITERIA

Patients will be a subset of patients participating in the multicenter IVUS protocol.

Willingness to travel to the NIH to participate in the NHLBI MRI/IMT study.

EXCLUSION CRITERIA

Pacemaker

Defibrillator

Brain aneurysm clips

Implanted active medical devices (neural stimulators, cochlear implants, insulin pumps, etc.)

Severe claustrophobia

Allergy to gadolinium based contrast agents (only excludes the gadolinium portion of the test)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125
Dates: Start 2004-04; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Corti R, Fuster V, Fayad ZA, Worthley SG, Helft G, Smith D, Weinberger J, Wentzel J, Mizsei G, Mercuri M, Badimon JJ. Lipid lowering by simvastatin induces regression of human atherosclerotic lesions: two years' follow-up by high-resolution noninvasive magnetic resonance imaging. Circulation. 2002 Dec 3;106(23):2884-7. doi: 10.1161/01.cir.0000041255.88750.f0. PMID 12460866
- [Background] Fayad ZA. MR imaging for the noninvasive assessment of atherothrombotic plaques. Magn Reson Imaging Clin N Am. 2003 Feb;11(1):101-13. doi: 10.1016/s1064-9689(02)00023-5. PMID 12797513
- [Background] Wasserman BA, Smith WI, Trout HH 3rd, Cannon RO 3rd, Balaban RS, Arai AE. Carotid artery atherosclerosis: in vivo morphologic characterization with gadolinium-enhanced double-oblique MR imaging initial results. Radiology. 2002 May;223(2):566-73. doi: 10.1148/radiol.2232010659. PMID 11997569